CLINICAL TRIAL: NCT01033188
Title: Single Bundle or Double Bundle Anterior Cruciate Ligament Reconstruction. A Randomized, Controlled Trial.
Brief Title: Double Bundle Anterior Cruciate Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Engebretsen, Professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6.2009.234
Record Dates: First submitted 2009-12-15; First posted 2009-12-16 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Knee Outcome, Subjective
Keywords: double bundle; hamstring graft; ACL reconstruction; single bundle

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Single-bundle technique (Active Comparator): Anatomic single-bundle technique
  Interventions: Procedure: Single bundle
- Double-bundle technique (Active Comparator): Anatomic double bundle technique
  Interventions: Procedure: Double bundle

INTERVENTIONS:
Procedure: Single bundle — Procedure:
  Transarthroscopic technique with medial portal placement of the femoral tunnel. Harvest of the semitendinosus/gracilis (ST/G) tendons through a 3-5 cm incision at the pes anserinus. The femoral tunnel is positioned at the anatomic foot print determined by the anatomic landmarks. The graft will be fixed with an Endobutton CL on the femur and with an Biosure PK screw in the tibia with the knee close to extension. Prior to the final fixation, the knee will be taken through flexion and extension movements.The surgery will be carried out by an experienced knee surgeon.
  Other Names: Endobutton
  Arms: Single-bundle technique
Procedure: Double bundle — Procedure:
  Transarthroscopic technique. Harvest of the semitendinosus/gracilis (ST/G) tendons through a 3-5 cm incision at the pes anserinus.Through a medial portal 2 tunnels will be anatomically placed in the foot print on the femur and the two tibial tunnels will be placed using the Smith & Nephew drill guide. The graft will be fixed with 2 Endobuttons on the femur and with 2 Biosure PK screws in the tibia. Prior to the final fixation, the knee will be taken through 20 flexion and extension movements. The PL bundle will be fixed with the knee close to ful extension. The surgery will be carried out by an experienced knee surgeon.
  Other Names: Endobutton
  Arms: Double-bundle technique

SUMMARY:
There has been an increased awareness towards ACL (anterior cruciate ligament) injuries for Norwegian teams, particularly in handball and soccer. The reported number of reconstructions in Norway ranges from 1500 to 2000 per year, and in the United States from 50,000 to 100,000 per year, making ACL reconstruction one of the most common orthopaedic procedures performed, especially among young, active and healthy individuals. However, reports state that there is a subset of patients (10-40%) who remain subjectively and objectively unstable and/or are unable to regain prior function. Additionally, it has been reported that degenerative joint disease is associated with traditional single-bundle ACL reconstructions in up to 50% of the patients in long term follow up studies.

It is well known that the ACL is composed of 2 functional bundles named after their tibial attachments, the anteromedial (AM) and posterolateral (PL) bundles.

It is believed that the current single-graft, single-bundle technique for reconstructing the anterior cruciate ligament does not anatomically reconstruct either one of these bundles.

In the last two years, the double bundle technique has been introduced and a few clinical studies are available, however only a few RCTs.

Further study is very important to determine if double-bundle ACL reconstructions should be performed, if single-bundle reconstructions can be adjusted to better adapt to their biomechanical insufficiency in restoring internal rotation torques and valgus moments, and also in trying to identify which patients might better benefit from single-bundle versus double-bundle ACL reconstructions.

DETAILED DESCRIPTION:
The aim of this study:

The primary aim is to compare the two operational techniques: single bundle hamstrings versus double bundle hamstrings ACL reconstruction, using the KOOS (Knee Osteoarthritis Outcome Score) Quality of Life(QoL) subscore as the primary outcome and clinical examinations, functional tests and standing radiographs (Kellgren Lawrence method) as secondary outcome measurements. Those assesments will be measured after 1,2 and 5 years after the operation.

Hypothesis:

There are no difference between the two methods as judged by the KOOS QoL subscore.

Questions to be answered:

Is there a difference between double-bundle and single-bundle technique in the subjective outcome scores as measured by the KOOS score? Are there differences between hamstrings single bundle and double bundle technique when the Lachman test and the pivot shift test are being used? Is there a difference between hamstrings double-bundle technique and single-bundle technique in return to sports and activity level? Are there differences between double-bundle technique and single -bundle technique in functional tests (one-leg hop test)? Is there a difference in the development of osteoarthritis between the two techniques?

ELIGIBILITY:
Inclusion Criteria:

* Clinically verified ACL rupture (history, Lachman test 2+ or more with no endpoint; pos pivot shift and arthroscopically verified) The graft used for AM bundle has a minimum size of 6.0 mm and 5.0 mm for t he PL bundle.

Exclusion Criteria:

* PCL injury,
* ACL injury to the contra lateral knee
* > 1+ medial or lateral-posterolateral ligament instability at operation date
* Previous ACL reconstruction
* Meniscal injury leaving < 50% of the meniscus intact
* Established OA as judged by Kellgren 3-4.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
KOOS score(QOL) | 1-5 years

SECONDARY OUTCOMES:
Standing radiographs (Kellgren Lawrence methode) | 3-5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Engebretsen, Phd, MD, Study Chair — Supervisor
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Aga C, Risberg MA, Fagerland MW, Johansen S, Troan I, Heir S, Engebretsen L. No Difference in the KOOS Quality of Life Subscore Between Anatomic Double-Bundle and Anatomic Single-Bundle Anterior Cruciate Ligament Reconstruction of the Knee: A Prospective Randomized Controlled Trial With 2 Years' Follow-up. Am J Sports Med. 2018 Aug;46(10):2341-2354. doi: 10.1177/0363546518782454. Epub 2018 Jul 18. PMID 30021073

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT01033188/SAP_000.pdf